CLINICAL TRIAL: NCT03357679
Title: Comparison of Bed up Head Elevated Intubation Position With Glidescope Assisted Tracheal Intubation: A Randomised, Controlled, Non-inferiority Trial
Brief Title: Comparison of Bed up Head Elevated Intubation Position With Glidescope Assisted Tracheal Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Samuel E H Tsan, MD, BMedSc, Doctor, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017112-5770
Record Dates: First submitted 2017-11-17; First posted 2017-11-30 (Actual); Last update posted 2018-09-17 (Actual); Status verified 2018-09

CONDITIONS: Bed up Head Elevated Intubation Position
Keywords: Bed up head elevated position; Glidescope assisted tracheal intubation; Laryngeal exposure; Time to intubation
MeSH Terms: interventions — Intubation, Intratracheal

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Investigator is blinded to the initial laryngeal exposure during the sniffing position, but is unblinded during assessment of laryngeal exposure in either the bed up head elevated position or glidescope assisted tracheal intubation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bed up head elevated intubation (Active Comparator): Patients positioned in the bed up head elevated position, followed by tracheal intubation
  Interventions: Procedure: Tracheal intubation; Device: Bed up head elevated tracheal intubation
- Glidescope assisted intubation (Active Comparator): Glidescope is used for laryngoscopy, followed by intubation
  Interventions: Procedure: Tracheal intubation; Device: Glidescope assisted tracheal intubation

INTERVENTIONS:
Procedure: Tracheal intubation — Intubation of the trachea with endotracheal tube
Device: Glidescope assisted tracheal intubation — With the use of the Glidescope video laryngoscope, the trachea will be intubated with the endotracheal tube
  Arms: Glidescope assisted intubation
Device: Bed up head elevated tracheal intubation — Use of the Macintosh laryngoscope blade size 3
  Arms: Bed up head elevated intubation

SUMMARY:
Positioning during the process of tracheal intubation is critical, as optimal positioning can greatly facilitate successful intubation. Many complications can occur as a result of failed intubation, ranging from airway injury, lack of oxygen, with even deaths. Today, the most popular positioning of patients for intubation is in the "sniffing" position. There is however evidence to support that intubation in the bed-up-head-elevated position may be better. In today's technological age, video assisted laryngoscopy (Laryngoscopy is the process of visualizing the vocal cords prior to intubation), a new method where the anaesthetist intubates a patient via aid of an image guided view of the airway, is increasingly popular due to its reliability and superiority to normal intubation. However, it is not widely available, and may suffer from technical breakdowns. The Glidescope is one example of a video laryngoscope, and has been widely researched in the medical literature. In this study, the investigators wish to investigate whether intubation in the bed-up-head-elevated position will be as good as, if not better than Glidescope assisted tracheal intubation, in patients undergoing elective surgery and planned for general anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing elective surgeries under general anaesthesia
2. Patients aged from 18 years old to 75 years old
3. Patients who are able to give informed consent

Exclusion Criteria:

1. Patients with airway obstruction
2. Patients with contraindications to neck extension
3. Patients with small mouth opening (<3 cm)
4. BMI > 35 kg/m3
5. Patients with ischemic heart disease, cerebrovascular disease and respiratory diseases
6. Patients in whom rapid sequence induction is indicated

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2017-12-26 (Actual); Primary Completion 2018-09-13 (Actual); Study Completion 2018-09-13 (Actual)

PRIMARY OUTCOMES:
Laryngeal exposure | Through study completion, period of 1 year
  Measured by Percentage of Glottic Opening (POGO) score. A 100% POGO score refers to visualisation of the entire glottic opening from the anterior commissure of the vocal cords to the interarytenoid notch. A POGO score of 0% refers to no visualisation of laryngeal structures. A 100% score is optimal.
Time required for intubation | Through study completion, period of 1 year
  Measured from the time the tip of the laryngoscope passes through the incisors to the time of the first recorded wave of capnography

SECONDARY OUTCOMES:
Number of intubation attempts | Through study completion, period of 1 year
Effort during laryngoscopy | Through study completion, period of 1 year
  Assessed based on a visual analogue scale, with 10 being the strongest effort, and 1 being the least effort required.
Complications arising from intubation | Through study completion, period of 1 year
  Incidence of hypoxia, hypotension, or esophageal intubation. Yes/no categories.
Airway trauma | Through study completion, period of 1 year
  Whether injury occurs to the lips, tongue, teeth, and other structures in the oropharyngeal area. Yes/no categories.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel E H Tsan, MD, BMedSc, Principal Investigator — University of Malaya
Locations (1):
- University Malaya Medical Centre, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tsan SEH, Lim SM, Abidin MFZ, Ganesh S, Wang CY. Comparison of Macintosh Laryngoscopy in Bed-up-Head-Elevated Position With GlideScope Laryngoscopy: A Randomized, Controlled, Noninferiority Trial. Anesth Analg. 2020 Jul;131(1):210-219. doi: 10.1213/ANE.0000000000004349. PMID 31348051